CLINICAL TRIAL: NCT00983320
Title: Quetiapine (Seroquel XR) for the Treatment of Fibromyalgia: a Clinical and Mechanistic Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Serge Marchand, PhD, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1443C00017
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; pain; quetiapine; randomized placebo controlled trial
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- medication (Experimental): quetiapine
  Interventions: Drug: quetiapine
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: quetiapine — flexible dosage (50 to 300 mg)
  Other Names: Seroquel XR
  Arms: medication
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled trial measuring the impact of quetiapine on clinical and experimental measures of pain in fibromyalgia and its biochemical correlates.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled trial measuring the impact of quetiapine on clinical and experimental measures of pain in fibromyalgia. The study also seeks to measure the hormonal, immunological and neurochemical correlates of clinical changes in time.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* A diagnosis of Fibromyalgia using the American College of Rheumatology criteria
* Females aged between 18 to 65 years
* Patients with an unsatisfactory response to their previous pharmacological treatment, defined as a score ≥4 on the pain severity item of the Fibromyalgia Impact Questionnaire
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment
* Patients receiving pharmacological treatment for fibromyalgia
* Able to understand and comply with the requirements of the study

Exclusion Criteria:

* Pregnancy or lactation
* Patients with DSM-IV Axis 1 disorder other than MDD and Chronic Pain Disorder within 6 months of enrolment
* Elderly patients with dementia and behavioural disturbances
* Patients who, in the investigator's opinion, pose a risk for suicide
* Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Patients already receiving an antipsychotic medication
* Current substance abuse/dependence (last year), as defined by DSM-IV criteria. Psychoactive substances include: alcohol, amphetamine, barbiturate, benzodiazepine, cannabis, cocaine, hallucinogen, opiates and phencyclidine
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment This could relate to patients with GI problems (short GI transit), Crohn's disease or disease requiring treatment with restricted medications as indicated in exclusion criteria items 5 and 6.
* Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension, hypotension) as judged by the investigator, based on the results from the physical exam, ECG, haematology, chemistry and urine screenings
* Participation in another drug trial within 4 weeks prior enrolment into this study
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

  * Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%.
  * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
  * Not under physician care for DM
  * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
  * Physician responsible for patient's DM care has not approved patient's participation in the study
  * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomization. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
  * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
* An absolute neutrophil count (ANC) of less or equal to 1.5 x 109 per liter

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia impact questionnaire | 12 weeks

SECONDARY OUTCOMES:
Thermal pain threshold | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Serge Marchand, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- University of Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] Hidalgo J, Rico-Villademoros F, Calandre EP. An open-label study of quetiapine in the treatment of fibromyalgia. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jan 30;31(1):71-7. doi: 10.1016/j.pnpbp.2006.06.023. Epub 2006 Aug 4. PMID 16889882